CLINICAL TRIAL: NCT03583073
Title: Reducing the Duration of Untreated Illness Among Youth in the Juvenile Justice System With Psychosis-Spectrum Disorders
Brief Title: Psychosis Screening in Juvenile Justice
Acronym: JJ-Psychosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Anthony Spirito, Professor, Brown University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: R34MH115457 (NIH); 1R34MH115457-01A1 (NIH)
Record Dates: First submitted 2018-06-28; First posted 2018-07-11 (Actual); Results first posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Psychotic Disorders; Psychosis Nos/Other
Keywords: psychosis; clinical high risk
MeSH Terms: conditions — Psychotic Disorders | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: The intervention will have two phases: 1) a Standard Care (baseline control) condition, followed by, 2) an Enhanced Referral/Linkage to Care condition. Because this is a roll-out trial, the two conditions will be compared using a non-randomized open trial design.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care/Baseline Control (Active Comparator): Standard care is the typical process of referral to mental health services for Juvenile Justice (JJ) youth who screen positive for mental heath concerns at intake. For this study, baseline control participants will be referred to the Coordinated Specialty Care (CSC) clinic due to their endorsement of psychosis-spectrum symptoms.
  Interventions: Behavioral: Standard Care
- Enhanced Referral/Linkage to Care (Experimental): The experimental condition will include a psychoeducational and motivational enhancement protocol completed at the JJS intake appointment, paired with a "warm hand-off" referral to the CSC for evaluation and initiation of mental health services.
  Interventions: Behavioral: Enhanced Referral/Linkage to Care

INTERVENTIONS:
Behavioral: Enhanced Referral/Linkage to Care — The JJ worker reviews with the family psychoeducation material about the role of mental health care in emotional/behavioral problems. The JJ intake worker will contact the CSC program directly with the family for a "warm hand-off". The CSC worker will speak with the parent and arrange for an intake evaluation. For families already receiving treatment, the CSC referral will be for consultation. Via phone, the CSC clinician will use a motivational interviewing style to encourage families to attend the appointment. Three and seven days after referral, the JJ worker will text the caregiver to see if the CSC appointment was kept. If not, the JJ worker will text the parent the CSC phone number and also ask permission to contact the CSC to assist the family in setting up another appointment.
  Arms: Enhanced Referral/Linkage to Care
Behavioral: Standard Care — Referral to the Coordinated Specialty Care (CSC) clinic
  Arms: Standard Care/Baseline Control

SUMMARY:
This study will investigate the occurrence of psychosis-spectrum disorders among youth in the Juvenile Justice System and track mental health referrals for these youth in Phase 1, a standard care condition. Then, in Phase 2, an enhanced referral and linkage to care model will be employed, with the aim of bolstering motivation for and engagement in mental health treatment. It is hypothesized that the enhanced referral protocol will promote completion of mental health care referrals.

DETAILED DESCRIPTION:
Among adolescents in the Juvenile Justice System (JJS), an estimated 3% have a psychotic illness, and it can be reasonably assumed that many more experience subthreshold psychotic-spectrum symptoms that may be indicative of risk. Evidence suggests that as many as 25% of those with first episode psychosis (FEP) have their first contact with care through criminal justice agencies. Duration of untreated psychosis (DUP), a negative prognostic factor, has been shown to be longer among those within the criminal justice system. This suggests that youth with psychotic symptoms who end up in the JJS may not receive appropriate mental health care. This study will first track mental health referrals for JJ youth with psychosis-spectrum symptoms in Phase 1, a standard care condition, and then an enhanced referral and linkage to care model will be investigated in Phase 2 of the study.

The current study will be conducted in the Rhode Island Family Court Juvenile Intake Department where all youth receive a mental health screen (Massachusetts Youth Screening Instrument - 2nd Ed; MAYSI -2). All youth who screen positive on the MAYSI-2 Thought Disturbance scale, and a second gate screening with the Prodromal Questionnaire - Brief Version (PQ-B), will be given referral information for Coordinated Specialty Care (CSC) services by JJS staff. Enrolled families will also participate in the research assessment, regardless of whether they pursue the CSC referral, which involves the Structured Interview for Psychosis-risk Syndromes [SIPS] and other measures to thoroughly assess history of psychotic symptoms, comorbid difficulties, and mental health care engagement. A comparison sample of youth who screen negative on the MAYSI-2 Thought Disturbance subscale will also be assessed with the SIPS to determine accuracy of the MAYSI-2/PQ-B screen in the identification of psychosis-risk. During the first phase of the study, JJS staff will follow standard procedures in referring youth to the state CSC. In the second phase of the study, JJS will be instructed in an enhanced referral/linkage to care protocol, including a "warm hand-off" where referrals will be put in direct and immediate contact with CSC staff. CSC staff will also be trained in procedures to increase the likelihood of follow through with the referral to the CSC. Three month follow-up qualitative interviews and quantitative assessments regarding referral pathways, bottlenecks and gaps in care, youth psychiatric symptoms, and JJS contacts will be conducted. This design maps onto the stated goals of PAR 16- 264 including: 1) Identify baseline rates of DUP within the JJS (and the investigators will also look at rates of psychosis-spectrum symptoms and disorders); 2) Map referral pathways to CSC; 3) Identify implementation and service level factors that create bottlenecks and gaps in linkage to the CSC; 4) Investigate the relationship between treatment linkage and psychotic symptoms/DUP; and, 5) Pilot test feasible strategies for reducing DUP.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent being seen in the Juvenile Justice System
* Legal guardian available to consent for juvenile's participation
* Adolescent assents to participate
* Adolescent is English speaking
* Parent/guardian may be English or Spanish-speaking
* Adolescent flags positive on the MAYSI-2 Thought Disturbance subscale or the PQ-B

Exclusion Criteria:

* Adolescent has observable developmental delays that would interfere with obtaining assent and/or accurate assessment
* Adolescent meets hospital level of care for imminent risk due to severity of symptoms

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 77 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Spirito, PhD, Principal Investigator — Brown University
Locations (2):
- United States (2):
  - Rhode Island Family Court, Providence, Rhode Island
  - Brown University, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 77 participants who screened positive for psychosis risk agreed to participate in the study.
Period: Overall Study
Arm/Group | Standard Care/Baseline Control | Enhanced Referral/Linkage to Care
Started | 45 | 32
Completed | 37 | 20
Not Completed | 8 | 12
Not completed — Lost to Follow-up | 8 | 12

BASELINE CHARACTERISTICS:
Population: There were 57 participants who screened positive for psychosis risk.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Care/Baseline Control | Enhanced Referral/Linkage to Care | Total
Number analyzed (Participants) | 37 | 20 | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 36 | 19 | 55
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.76 (1.53) | 14.30 (1.56) | 14.60 (1.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 13 | 31
  Male | 19 | 7 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 6 | 19
  White | 16 | 12 | 28
  More than one race | 5 | 2 | 7
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 37 | 20 | 57

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Used Outpatient Mental Health Services
Description: Number of Participants who Used Any Outpatient Mental Health Services by Participant's Caregiver Report
Time Frame: 3-month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care/Baseline Control | Enhanced Referral/Linkage to Care
Number analyzed (Participants) | 37 | 20
Participants | 20 | 9
Statistical Analysis 1: Comparison: Standard Care/Baseline Control vs Enhanced Referral/Linkage to Care; Test type: Superiority; p = .053, Chi-squared, Corrected; DF = 1

2. Secondary Outcome: Psychosis-spectrum Positive Symptoms
Description: Psychosis-spectrum subscale of The Structured Interview for Psychosis-risk Syndromes (SIPS) has five positive symptoms including odd or delusional thoughts, paranoia/suspiciousness, grandiosity, perceptual abnormalities, and disorganized communication. Each symptom is scored on a scale from 0 to 6 and a total suscale score is calculated, ranging from 0 to 30. Higher scores indicate greater severity of positive symptoms and potentially higher risk for developing psychosis.
Time Frame: 3-month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Care/Baseline Control | Enhanced Referral/Linkage to Care
Number analyzed (Participants) | 37 | 20
score on a scale | 5.89 (3.64) | 3.95 (4.12)
Statistical Analysis 1: Comparison: Standard Care/Baseline Control vs Enhanced Referral/Linkage to Care; Test type: Superiority; p = .072, Chi-squared, Corrected; Mean Difference (Final Values) = 1.94, 95% CI 2-sided [-0.18 to 4.06]

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Standard Care/Baseline Control | Enhanced Referral/Linkage to Care
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/20
Other Adverse Events (participants affected / at risk) | 0/37 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-09-01): https://cdn.clinicaltrials.gov/large-docs/73/NCT03583073/Prot_SAP_001.pdf
  • Informed Consent Form (2020-03-13): https://cdn.clinicaltrials.gov/large-docs/73/NCT03583073/ICF_002.pdf